CLINICAL TRIAL: NCT07280182
Title: Comparing the Early Postoperative Analgesic Effect of the Transmuscular Quadratus Lumborum Block Versus the Lumbar Plexus Block for Patients Undergoing Spiral Thighplasty Surgery
Brief Title: Effect of the Quadratus Lumborum Block Versus the Lumbar Plexus for Spiral Thighplasty Surgery
Acronym: QLB&LPB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Amal Gouda Elsayed Safan, lecturer, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 11/2025ANET2; Menoufia University (Registry Identifier: Faculty of medicine)
Record Dates: First submitted 2025-11-28; First posted 2025-12-12 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Analgesia
Keywords: spiral thighplasty , pain , nerve block
MeSH Terms: conditions — Agnosia; Pain | interventions — Dental Occlusion

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, parallel-group, double-blind, clinical trial. Primary endpoint: time for first analgesic request postoperatively. Key secondary endpoints: 24-hour opioid consumption (oral morphine equivalents), pain on movement at 6/12/24 hours, time to first ambulation, postoperative nausea/vomiting (PONV), block performance time, and block-related complications. Hypothesis: QLB is non-inferior to LPB for 24-hour pain scores and will yield less motor weakness
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Computer-generated randomization in variable blocks; allocation sealed in opaque envelopes. Blocks performed by an anesthesiologist not involved in postoperative assessment. Patients and outcome assessors are blinded. Drape and opaque dressings conceal injection sites for both groups to preserve blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group QLB (Other): Ultrasound-Guided Trans-muscular QLB
  Interventions: Other: Ultrasound-Guided Trans-muscular QLB
- Group LPB (Other): Ultrasound-Guided Posterior Lumbar Plexus (Psoas Compartment) Block
  Interventions: Other: Ultrasound-Guided Posterior Lumbar Plexus (Psoas Compartment) Block

INTERVENTIONS:
Other: Ultrasound-Guided Trans-muscular QLB — With the patient lateral decubitus position, a low-frequency curvilinear probe in the 'Shamrock' view at L2-L4. In-plane posterior-to-anterior needle advancement through the Quadratus lumborum to the interfascial plane anterior to QL and posterior to Psoas major. Inject 30 mL Bupivacaine 0.25% after negative aspiration and hydrodissection to confirm proper spread . Then the patient will be turned to the other side, and the block will be done with the same technique
  Arms: Group QLB
Other: Ultrasound-Guided Posterior Lumbar Plexus (Psoas Compartment) Block — Lateral decubitus, Shamrock view to identify the Psoas compartment; in-plane needle advancement to the Psoas compartment adjacent to the transverse process. Inject 30 mL of Bupivacaine 0.25% in 5 mL increments, aspirating frequently. This will be done in the same position for both sides
  Arms: Group LPB

SUMMARY:
Whether trans muscular QLB provides postoperative analgesia compared with LPB after thigh lift surgery

DETAILED DESCRIPTION:
Adequate analgesia after spiral thigh reduction (thigh lift) is essential for early mobilization and patient satisfaction. Quadratus lumborum block (QLB) has shown analgesic efficacy comparable to lumbar plexus block (LPB) for hip area surgery with potential advantages in motor-sparing and safety

ELIGIBILITY:
Inclusion Criteria:

* ASA ( American Society of Anaesthesia) I-II
* elective bilateral spiral thigh lift under general anesthesia
* consent to regional block and trial participation

Exclusion Criteria:

* Coagulopathy or therapeutic anticoagulation not meeting ASRA safety windows
* infection at injection sites
* allergy to local anesthetics
* preexisting significant neuropathy
* BMI > 35 kg/m² if impeding ultrasound visualization; renal/hepatic failure; pregnancy; inability to use NRS; chronic opioid use >60 mg oral morphine equivalents/day; contraindication to study analgesics.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2025-11-27 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale score | 24 hours
  Visual analogue scale score at 1st,6th,12th and 24 h (where 0 is interpreted as no pain, 1-4 mild pain, 5-6 moderate pain, 7-10 severe pain)

SECONDARY OUTCOMES:
Time for first analgesic request | 24 hours
  first analgesic request
Opioid consumption | 24 hours
  cumulative opioid consumption
Time to walk >30 (meter) | 24 hours
  walk >30 (meter)
Performance Time | minutes
  block performance time
The number of patients who develop block-related complications | 24 hours
  nausea and vomiting , hypotension
the patients Satisfaction questionnaire | 24 hours
  pateints are either : Dissatisfied Neither satisfied nor dissatisfied Satisfied Very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: AMAL G SAFAN, MD, Study Director — Menoufia University
Locations (1):
- Faculty of medicine,Menofia university hospitals, Cairo, Shibin El Kom, Egypt

IPD SHARING:
Plan to Share IPD: No